CLINICAL TRIAL: NCT03585140
Title: Effect of Adding a Diet With Low Glycemic Index and Load During 12 Weeks for the Treatment of Moderate Acne in Adults: a Randomized Clinical Trial
Brief Title: Low Glycemic Index and Load Diet for the Treatment of Acne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Dermatológico Dr. Ladislao de la Pascua (Other)
Responsible Party: Principal Investigator, Dra. Martha Alejandra Morales Sánchez, MD, Centro Dermatológico Dr. Ladislao de la Pascua
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 106/2016
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Acne Vulgaris; Diet Modification
Keywords: Acne Vulgaris; Low Glycemic Diet; Doxycycline; Adapalene
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Gels; Doxycycline

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial, two-arm
Who Masked: Investigator, Outcomes Assessor
Masking Description: Diet intervention was made by the nutrition specialist. Neither the principal investigator nor the outcome assessor were aware about the group of diet intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Diet (Active Comparator): Participants will receive a normal diet according to their metabolic status.
  Interventions: Other: Normal diet; Drug: Adapalene 0.1% Gel; Drug: Doxycycline
- Low glycemic diet (Experimental): Participants will receive a low-glycemic index and load diet according to their metabolic status. Milk and vitamin supplements will be eliminated from the diet.
  Interventions: Other: Low glycemic diet; Drug: Adapalene 0.1% Gel; Drug: Doxycycline

INTERVENTIONS:
Other: Normal diet — The energy consumption of each of the participants will be calculated, using the Mifflin-St Jeor formula. Each participant will receive a standard menu of 6 days according to their metabolic requirements and a list of equivalent foods. The distribution of macronutrients will be: 45% carbohydrates, 30% lipids and 25% proteins.
  Arms: Normal Diet
Other: Low glycemic diet — The energy consumption of each of the participants will be calculated, using the Mifflin-St Jeor formula. Each participant will receive a standard menu of 6 days according to their metabolic requirements and a list of equivalent foods. A list of foods classified as having low index and glycemic load was used according to the mexican equivalent food system. The distribution of macronutrients will be: 45% carbohydrates, 30% lipids and 25% proteins. Milk and vitamin supplements will be eliminated from the diet.
  Arms: Low glycemic diet
Drug: Adapalene 0.1% Gel — Adapalene 0.1% gel daily at night for 12 weeks, applied on the face, chest and back.
  Other Names: Adapalene
Drug: Doxycycline — Doxycycline 100 mg per day orally, before breakfast

SUMMARY:
Clinical trial to determine the effect of adding a diet with low glycemic index and load to adults for the treatment of moderate acne. Adult patients with acne where recruited in two groups, A and B. Group A received a normal diet according to their metabolic status and group B received a diet with low glycemic index and load. Outcomes were measured at week 12.

DETAILED DESCRIPTION:
Clinical trial to determine the effect of adding a diet with low glycemic index and load to adults for the treatment of moderate acne. Adult patients with acne where recruited in two groups, A and B. Both groups of treatment were treated with doxycycline 100 mg per day plus adapalene 0.1% gel daily for 12 weeks. During pharmacologic treatment, all patients had nutrition counseling monthly. Group A received a normal diet according to their metabolic status and group B received a diet with low glycemic index and load. At the end of the trial, the change in acne lesions count was analyzed and also their metabolic status. Quality of life was also measured.

ELIGIBILITY:
Inclusion Criteria:

* Having moderate inflammatory acne
* 18 to 25 years old
* Male
* Stable weight during the last 3 months

Exclusion Criteria:

* Previous or actual isotretinoin therapy
* Antibiotic therapy or during the last 3 months
* Therapy based on peelings, dermabrasion, laser or intense pulsed light during the last 6 months
* Endocrine disorders
* Drug and alcohol consumption during the last 6 months
* Tabacco use during the last 6 months
* Lactose intolerance
* Have eating disorders or gastrointestinal disorders
* Actual nutrition therapy
* Have chronic diseases that requires pharmacologic therapy
* Severe acne that requires isotretinoin therapy

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Count of inflammatory acne lesions | 12 weeks
  Number of papules and pustules

SECONDARY OUTCOMES:
Count of non-inflammatory acne lesions | 12 weeks
  Number of comedones
Changes in quality of life | 12 weeks
  Score of the Dermatology Life Quality Index

CONTACTS AND LOCATIONS:
Overall Officials: Martha A Morales-Sánchez, MD, Principal Investigator — Centro Dermatológico Dr. Ladislao de la Pascua